CLINICAL TRIAL: NCT03966170
Title: Efficacy of Citicoline as Neuroprotector in Preterm; A Randomized Controlled Trial
Brief Title: Citicoline as Neuroprotector in Preterm
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Citicoline
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Pre-Term
MeSH Terms: conditions — Premature Birth | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citicoline (Experimental): Citicoline as neuroprotector
  Interventions: Drug: Citicoline
- Placebo drug (Placebo Comparator): Placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Citicoline — Citicoline as neuroprotector
  Arms: Citicoline
Drug: Placebo oral tablet — placebo drug
  Arms: Placebo drug

SUMMARY:
Citicoline as neuroprotector in preterm

DETAILED DESCRIPTION:
Efficacy of Citicoline as neuroprotector in preterm; A randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Preterm on CPAP or ventilator

Exclusion Criteria:

* Multiple congenital anomalies

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of children with affection of the brain | 6 months
  Number of children with affection of the brain

CONTACTS AND LOCATIONS:
Overall Officials: May R Elsheikh, MD, Principal Investigator — Tanta University - Faculty of Medicine; Abeer Salamah, MD, Study Director — Kafr-Elsheikh University - Faculty of Medicine
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No